CLINICAL TRIAL: NCT02171585
Title: Relative Bioavailability of Dabigatran After Single Oral Administration of 150 mg Dabigatran Etexilate (Capsule) With or Without Multiple Oral Administration of 500 mg Clarithromycin (Tablet) Bid in Healthy Male and Female Volunteers (an Open Label, Fixed Sequence, Clinical Phase I Study)
Brief Title: Bioavailability of Dabigatran With or Without Clarithromycin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.82
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Clarithromycin

ARMS (2):
- Dabigatran without Clarithromycin (Experimental)
  Interventions: Drug: Dabigatran etexilate
- Dabigatran with Clarithromycin (Experimental)
  Interventions: Drug: Dabigatran etexilate; Drug: Clarithromycin

INTERVENTIONS:
Drug: Dabigatran etexilate
Drug: Clarithromycin
  Arms: Dabigatran with Clarithromycin

SUMMARY:
To investigate whether and to what extent the reported potent P-gp inhibitor clarithromycin affects pharmacokinetic parameters (area under the curve (AUC) and maximal concentration (Cmax)) of dabigatran.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females ≥18 and ≤50 years of age, based on a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests.
* Body mass index (BMI) ranging from 18.5 to 29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsade de Pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)
* In addition, the following exclusion criteria applied to females:

  * Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
  * No adequate contraception during the study and until 1 month of study completion, (implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence [for at least 1 month prior to enrolment], vasectomised partner [vasectomy performed at least 1 year prior to enrolment], or surgical sterilisation [including hysterectomy] were considered adequate contraception. Females whose partner was not vasectomised, were not sexually abstinent, or surgically sterile were asked to use barrier contraception methods (e.g. condom, diaphragm with spermicide)
  * Lactation period
* Intake of medication, which influenced blood coagulation, including acetylsalicylic acid and oral vitamin K antagonists, among others

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ of total dabigatran (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
Cmax of total dabigatran (maximum measured concentration of the analyte in plasma) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5

SECONDARY OUTCOMES:
AUC0-∞ of free dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
Cmax of free dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
Cmax of clarithromycin | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
AUC0-12 of clarithromycin (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 12 h) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
AUC0-tz of clarythromycin (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
AUCτ,1 of clarythromycin (area under the concentration time curve over one dosing interval after the first dose) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
AUC0-24 of clarythromycin (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 h after the administration) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
tmax of clarythromycin (time from dosing to the maximum concentration of the analyte in plasma) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
λz (terminal rate constant in plasma) of clarythromycin | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
t1/2 of clarythromycin (terminal half-life of the analyte in plasma) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
MRTpo of clarythromycin (mean residence time of the analyte in the body after oral administration) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
CL/F of clarythromycin (apparent clearance of the analyte in the plasma after extravascular administration) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
Vz/F of clarythromycin (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after first dose of clarythromycin on day 1 of visit 3
AUC0-tz of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
AUCτ,1 of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
AUC0-24 of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
tmax of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
λz of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
t1/2 of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
MRTpo of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
CL/F of dabigatran | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
Vz/F of dabigatran (free and total) | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34 hours after administration of study drug on day 1 of visits 2, 3, and 5
AUCτ,ss of clarythromycin (area under the concentration-time curve of the analyte in plasma within the uniform dosing interval τ) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
AUC0-tz,ss of clarythromycin (area under the concentration-time curve of the analyte in plasma from the time point 0 after the last dose at steady state to the last quantifiable analyte plasma concentration within the uniform dosing interval τ) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
Cmax,ss of clarythromycin (maximum concentration of the analyte in plasma at steady state) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
tz,ss of clarythromycin (time of last measurable concentration of the analyte in plasma within the dosing interval τ at steady state) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
tmax,ss of clarythromycin (time from last dosing to the maximum concentration of the analyte in plasma at steady state on day 4) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
CL/F,ss of clarythromycin (apparent clearance of the analyte in the plasma at steady state after extravascular multiple dose administration) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
Cmin,ss of clarythromycin (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
tmin,ss of clarythromycin (time from last dosing to the minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
Cpre,ss of clarythromycin (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
MRTpo,ss of clarythromycin (mean residence time of the analyte in the body at steady state after oral administration) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
Vz/F,ss of clarythromycin (apparent volume of distribution during the terminal phase λz at steady state following an extravascular administration) | Before and 30 min, 55 min, 1.5, 2, 2.5, 3, 4, 5, 7, 9, 11, 13, 25 hours after multiple dosing of clarythromycin on day 1 of visit 4 and 5
Ae0-24 of dabigatran (amount of analyte eliminated in urine from the time interval 0-24h) | Day 1 to 2 of visits 2, 3 and 5
fe0-24 of dabigatran (fraction of administered drug excreted unchanged in urine from time point 0-24h) | Day 1 to 2 of visits 2, 3 and 5
CLR, 0-24 of dabigatran (renal clearance of the analyte in plasma from the time point 0 until the time point 24h ) | Day 1 to 2 of visits 2, 3 and 5
Changes in thrombin time (TT) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours after administration of study drug on day 1 of visits 2, 3 and 5
Changes in ecarin clotting time (ECT) | 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours after administration of study drug on day 1 of visits 2, 3 and 5
Occurrence and intensity of adverse events | up to 21 days
Assessment of tolerability by investigator | Day 21
Changes from baseline in physical examination | Baseline, day 21
Changes in vital signs (blood pressure, pulse rate) | up to day 21
Changes in 12-lead electrocardiogram (ECG) | up to day 21
Changes in clinical laboratory tests | up to day 21